CLINICAL TRIAL: NCT02710370
Title: Intestinal Metabolic Reprogramming as a Key Mechanism of Gastric Bypass in Humans
Status: Active, not recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Harvard University (Other); National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Anita P. Courcoulas, Director, Minimally Invasive Bariatric & General Surgery, University of Pittsburgh
Other Study IDs: STUDY19060074; R01DK108642 (NIH)
Record Dates: First submitted 2016-02-05; First posted 2016-03-16 (Estimated); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Obesity; Diabetes Mellitus, Type 2; Endocrine System Diseases; Glucose Metabolism Disorders; Metabolic Diseases
Keywords: Bariatric Surgery; Gastric Bypass; Obesity/surgery; Endoscopy, Digestive System; Blood Glucose/metabolism; Diabetes Mellitus, Experimental/metabolism; Energy Metabolism; Glucose/metabolism; Jejunum/metabolism; Metabolomics; Gene Expression
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Endocrine System Diseases; Glucose Metabolism Disorders; Metabolic Diseases; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Intestinal samples, serum and plasma will be collected from patients who have had gastric bypass surgery. Tissue samples will be processed for histo-morphological examination and for RNA, protein and metabolomics analyses.
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- Controls: Patients who meet criteria for gastric bypass surgery, and do not have a documented history of Type 1 or Type 2 Diabetes.
- Participants with Type 2 Diabetes: Patients who meet criteria for gastric bypass surgery, and have a documented history of Type 2 Diabetes.

SUMMARY:
The purpose of this research study is to determine how gastric bypass surgery effects metabolism in obesity and Type 2 Diabetes. One mechanism that has been investigated in animal models is change to the biology of the small intestine (Roux limb) and how glucose and other fuels are metabolized (or how the body digests and uses sugar and other fuels). This study will evaluate the role of the intestine in the beneficial metabolic effects of gastric bypass surgery. It specifically will examine whether the intestine increases its metabolism and its activity, and whether this results in an increase in fuel utilization. Thirty two (32) subjects will be recruited (18 with and 14 without Type 2 Diabetes). At the time of gastric bypass surgery, a small piece of intestine that is usually discarded will be collected. At three time points over the first year after surgery, intestinal samples will be obtained by endoscopy or insertion of a lighted flexible tube through the mouth. Blood samples will be taken at all time points, as well. All samples will undergo comprehensive metabolic analyses. Comparisons will be made between the two groups to understand the metabolic changes over time and if there are differences between the two groups.

DETAILED DESCRIPTION:
Several studies have concluded that Roux-en-Y gastric bypass surgery (RYGBS) is the best current treatment option for obesity-related Type 2 Diabetes Mellitus (T2DM). The mechanisms underlying RYGBS-induced improvement in glycemic control remain unclear. Many investigators have advocated that this effect does not depend upon body weight loss, based on clinical observations that improvement in glucose homeostasis occurs early in the postoperative period, often prior to hospital discharge. Understanding the mechanisms underlying the metabolic effects of RYGBS will help to engineer ways to improve RYGB or to produce these effects without surgery.

This study will examine the concept of intestinal metabolic reprogramming as one of the key mechanisms of action for diabetes improvement following Roux-en-Y gastric bypass surgery (RYGBS) in humans. It is hypothesized that the reconfigured intestine is characterized by an increase in energetically expensive processes, such as structural remodeling, cytoskeletal reorganization, and cellular proliferation. To accommodate the increased bioenergetics demands, the intestinal epithelium increases its metabolic activity and reprograms its fuel utilization. Specifically, glucose, cholesterol and amino acid metabolism are all dramatically altered to increase anabolic pathways and generate building blocks for cellular growth and maintenance.

It has not previously been possible to test this hypothesis in humans as: A) the adaptive processes of the intestine in patients undergoing RYGBS have not been thoroughly characterized, B) it is not known whether the intestinal reprogramming appears early enough to explain the prompt improvement in glucose metabolism observed after RYGBS in humans, and C) the variability of the degree of intestinal metabolic adaptation, which could account for the variability in remission of T2DM, has not been studied. This study will perform a longitudinal, comprehensive metabolic analysis of the Roux limb in human subjects with and without T2DM undergoing RYGBS and determine the time course of the adaptive metabolic changes.

Eighteen (18) subjects with and fourteen (14) subjects without T2DM (total 32 subjects), who have been scheduled to undergo RYGBS as standard of care, will be recruited. For each enrolled subject, data collection will include an intestinal tissue sample (Roux limb tissue sampling from discarded tissue) at the time of RYGBS, from the mucosa of the jejunum, within 40 cm from the gastrojejunal anastomosis. Postoperatively, tissue sampling from the same area will be performed by an Upper GI endoscopy, at 1 month (±15 days), 6 months (±1 month) and 12 months (±2 months) after RYGBS. Tissue samples will be processed for histo-morphological examination and for RNA, protein and metabolomics analyses. A blood sample will be obtained at all time points and analyzed for metabolic biomarkers. Data analysis will include description and comparison of the morphological, gene protein and metabolite signatures of the intestinal (Roux limb) tissue and the blood biomarkers from each time point. Additionally, these outcome measures will be compared between the two groups (T2DM and Non-T2DM). Finally, a correlation of the intestinal adaptive changes with metabolic status, some eating behaviors, adverse symptomatology, and quality of life will be undertaken.

ELIGIBILITY:
Inclusion Criteria:

* Patients who elect to undergo gastric bypass surgery
* Standard bariatric surgery criteria (A BMI 35 to 40 kg/m2, with an obesity comorbid condition, OR BMI 40 kg/m2 or >).

Exclusion Criteria:

* Prior bariatric or foregut surgery
* Documented history of Type 1 Diabetes
* Poor overall general health
* Impaired mental status
* Drug and/or alcohol addiction
* Currently smoking
* Pregnant or plans to become pregnant
* Portal hypertension and/or cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who plan to undergo gastric bypass, with or without Type 2 Diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2016-02; Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Description of intestinal morphology. | Baseline, at time of operation
  Histology and electron microscopy will be used to assess cellular architecture, brush border, cytoskeleton and junctions, and the size and shape of organelles.
Description of intestinal morphology. | 1 month after surgery.
  Histology and electron microscopy will be used to assess cellular architecture, brush border, cytoskeleton and junctions, and the size and shape of organelles.
Description of intestinal morphology. | 6 months after surgery.
  Histology and electron microscopy will be used to assess cellular architecture, brush border, cytoskeleton and junctions, and the size and shape of organelles.
Description of intestinal morphology. | 12 months after surgery.
  Histology and electron microscopy will be used to assess cellular architecture, brush border, cytoskeleton and junctions, and the size and shape of organelles.
Characterization of gene and protein expression of markers of cellular proliferation, cytoskeletal remodeling, and cellular machinery of glucose and cholesterol metabolic pathways. | Baseline, at time of operation.
  Gene expression (RT-PCR) and protein expression (western blotting) for about 100 markers of cellular proliferation (e.g., cyclins, MKi67, PCNA), cytoskeletal remodeling (e.g., brush border enzymes and proteins), cellular machinery of glucose and cholesterol metabolic pathways (e.g., glucose transporters, enzymes of biochemical pathways).
Characterization of gene and protein expression of markers of cellular proliferation, cytoskeletal remodeling, and cellular machinery of glucose and cholesterol metabolic pathways. | 1 month after surgery.
  Gene expression (RT-PCR) and protein expression (western blotting) for about 100 markers of cellular proliferation (e.g., cyclins, MKi67, PCNA), cytoskeletal remodeling (e.g., brush border enzymes and proteins), cellular machinery of glucose and cholesterol metabolic pathways (e.g., glucose transporters, enzymes of biochemical pathways).
Characterization of gene and protein expression of markers of cellular proliferation, cytoskeletal remodeling, and cellular machinery of glucose and cholesterol metabolic pathways. | 6 months after surgery.
  Gene expression (RT-PCR) and protein expression (western blotting) for about 100 markers of cellular proliferation (e.g., cyclins, MKi67, PCNA), cytoskeletal remodeling (e.g., brush border enzymes and proteins), cellular machinery of glucose and cholesterol metabolic pathways (e.g., glucose transporters, enzymes of biochemical pathways).
Characterization of gene and protein expression of markers of cellular proliferation, cytoskeletal remodeling, and cellular machinery of glucose and cholesterol metabolic pathways. | 12 months after surgery.
  Gene expression (RT-PCR) and protein expression (western blotting) for about 100 markers of cellular proliferation (e.g., cyclins, MKi67, PCNA), cytoskeletal remodeling (e.g., brush border enzymes and proteins), cellular machinery of glucose and cholesterol metabolic pathways (e.g., glucose transporters, enzymes of biochemical pathways).
Description of metabolite profile of the intestine and serum/plasma. | Baseline, at time of operation.
  Metabolite profiling of the tissues and serum/plasma, using mass spectrometry techniques.
Description of metabolite profile of the intestine and serum/plasma. | 1 month after surgery.
  Metabolite profiling of the tissues and serum/plasma, using mass spectrometry techniques.
Description of metabolite profile of the intestine and serum/plasma. | 6 months after surgery.
  Metabolite profiling of the tissues and serum/plasma, using mass spectrometry techniques.
Description of metabolite profile of the intestine and serum/plasma. | 12 months after surgery.
  Metabolite profiling of the tissues and serum/plasma, using mass spectrometry techniques.
Change from baseline (time of operation) in morphological signatures. | Baseline (0 months) and 1 month, 6 months and 12 months post-surgery.
Change from baseline (time of operation) in gene and protein expression for markers of cellular proliferation, cytoskeletal remodeling, and cellular machinery of glucose and cholesterol metabolic pathways. | Baseline (0 months) and 1 month, 6 months and 12 months post-surgery.
Change from baseline (time of operation) in metabolite profile. | Baseline (0 months) and 1 month, 6 months and 12 months post-surgery.

SECONDARY OUTCOMES:
Comparison of intestinal morphology signature between patients with and without diabetes. | Baseline (0 months) and 1 month, 6 months and 12 months post-surgery.
Comparison of gene and protein expression profiles and levels of expression of markers of cellular proliferation, cytoskeletal remodeling, and cellular machinery of glucose and cholesterol metabolic pathways between patients with and without diabetes. | Baseline (0 months) and 1 month, 6 months and 12 months post-surgery.
Comparison of metabolite profile between patients with and without diabetes. | Baseline (0 months) and 1 month, 6 months and 12 months post-surgery.
Correlation of intestinal morphology signature with eating behaviors. Assessed by specific questionnaire. | Baseline (0 months) and 1 month, 6 months and 12 months post-surgery.
  Morphology as described in Primary Measures 1 - 4 correlated with eating behaviors as obtained and described by the Eating and Weight History Form (EWH).
Correlation of eating behaviors with gene and protein expression of markers of cellular proliferation, cytoskeletal remodeling, and cellular machinery of glucose and cholesterol metabolic pathways. Assessed by specific questionnaire. | Baseline (0 months) and 1 month, 6 months and 12 months post-surgery.
  Gene and protein expression of markers of cellular proliferation, cytoskeletal remodeling, and cellular machinery of glucose and cholesterol metabolic pathways as described in Primary Measures 5 - 8 correlated with eating behaviors as obtained and described by the Eating and Weight History Form (EWH).
Correlation of metabolite profile with eating behaviors. Assessed by specific questionnaire. | Baseline (0 months) and 1 month, 6 months and 12 months post-surgery.
  Intestinal and serum/plasma metabolite profiling as described in primary outcomes 9 - 12 correlated with eating behaviors as obtained and described by the Eating and Weight History Form (EWH).
Correlation of intestinal morphology signature with quality of life assessed by SF-36 Instrument. | Baseline (0 months) and 1 month, 6 months and 12 months post-surgery.
  Morphology as described in Primary Measures 1 - 4 correlated with quality of life as measured by the SF-36 Instrument (total and subscales).
Correlation of quality of life assessed by SF-36 Instrument with gene and protein expression for markers of cellular proliferation, cytoskeletal remodeling, and cellular machinery of glucose and cholesterol metabolic pathways. | Baseline (0 months) and 1 month, 6 months and 12 months post-surgery.
  Gene and protein expression of markers of cellular proliferation, cytoskeletal remodeling, and cellular machinery of glucose and cholesterol metabolic pathways as described in Primary Measures 5 - 8 correlated with quality of life as measured by the SF-36 Instrument (total and subscales).
Correlation of metabolite profile with quality of life assessed by SF-36 Instrument. | Baseline (0 months) and 1 month, 6 months and 12 months post-surgery.
  Intestinal and serum/plasma metabolite profiling as described in primary outcomes 9 - 12 correlated with quality of life as measured by the SF-36 Instrument (total and subscales).
Correlation of intestinal morphology signature with adverse symptomatology (e.g., Dumping syndrome, Hypoglycemia). Assessed by specific questionnaires. | Baseline (0 months) and 1 month, 6 months and 12 months post-surgery.
  Morphology as described in Primary Measures 1 - 4 correlated with dumping syndrome characteristics as defined on the Sigstad Clinical Diagnostic Index and the Gastrointestinal and Neurological Symptom Form and hypoglycemic symptoms as described on the Glycemic Symptom Form.
Correlation of adverse symptomatology (Dumping syndrome, Hypoglycemia) with gene/protein expression of markers of cellular proliferation, cytoskeletal remodeling, and cellular machinery of glucose and cholesterol metabolic pathways. | Baseline (0 months) and 1 month, 6 months and 12 months post-surgery.
  Gene and protein expression levels of markers of cellular proliferation, cytoskeletal remodeling, and cellular machinery of glucose and cholesterol metabolic pathways as described in Primary Measures 5 - 8 correlated with dumping syndrome characteristics as defined on the Sigstad Clinical Diagnostic Index and the Gastrointestinal and Neurological Symptom Form and hypoglycemic symptoms as described on the Glycemic Symptom Form.
Correlation of metabolite profile with adverse symptomatology (e.g., Dumping syndrome, Hypoglycemia). Assessed by specific questionnaires. | Baseline (0 months) and 1 month, 6 months and 12 months post-surgery.
  Intestinal and serum/plasma metabolite profiling as described in primary outcomes 9 - 12 correlated with dumping syndrome characteristics as defined on the Sigstad Clinical Diagnostic Index and the Gastrointestinal and Neurological Symptom Form and hypoglycemic symptoms as described on the Glycemic Symptom Form.
Generation of intestinal organoids from Roux limb biopsies. | Baseline (0 months) and 1 month, 6 months and 12 months post-surgery. We began collection in August 2017 on some participants.
  Feasibility of the generation of intestinal organoids for targeted mechanistic studies in vitro.

CONTACTS AND LOCATIONS:
Overall Officials: Anita Courcoulas, MD, MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Saeidi N, Meoli L, Nestoridi E, Gupta NK, Kvas S, Kucharczyk J, Bonab AA, Fischman AJ, Yarmush ML, Stylopoulos N. Reprogramming of intestinal glucose metabolism and glycemic control in rats after gastric bypass. Science. 2013 Jul 26;341(6144):406-10. doi: 10.1126/science.1235103. PMID 23888041
- [Background] Laferrere B. Do we really know why diabetes remits after gastric bypass surgery? Endocrine. 2011 Oct;40(2):162-7. doi: 10.1007/s12020-011-9514-x. Epub 2011 Aug 19. PMID 21853297
- [Background] Courcoulas AP, Christian NJ, Belle SH, Berk PD, Flum DR, Garcia L, Horlick M, Kalarchian MA, King WC, Mitchell JE, Patterson EJ, Pender JR, Pomp A, Pories WJ, Thirlby RC, Yanovski SZ, Wolfe BM; Longitudinal Assessment of Bariatric Surgery (LABS) Consortium. Weight change and health outcomes at 3 years after bariatric surgery among individuals with severe obesity. JAMA. 2013 Dec 11;310(22):2416-25. doi: 10.1001/jama.2013.280928. PMID 24189773
- [Background] Stylopoulos N, Hoppin AG, Kaplan LM. Roux-en-Y gastric bypass enhances energy expenditure and extends lifespan in diet-induced obese rats. Obesity (Silver Spring). 2009 Oct;17(10):1839-47. doi: 10.1038/oby.2009.207. Epub 2009 Jun 25. PMID 19556976
- [Background] Arterburn DE, Courcoulas AP. Bariatric surgery for obesity and metabolic conditions in adults. BMJ. 2014 Aug 27;349:g3961. doi: 10.1136/bmj.g3961. PMID 25164369
- [Background] Nestoridi E, Kvas S, Kucharczyk J, Stylopoulos N. Resting energy expenditure and energetic cost of feeding are augmented after Roux-en-Y gastric bypass in obese mice. Endocrinology. 2012 May;153(5):2234-44. doi: 10.1210/en.2011-2041. Epub 2012 Mar 13. PMID 22416083
- [Background] Stefater-Richards MA, Panciotti C, Feldman HA, Gourash WF, Shirley E, Hutchinson JN, Golick L, Park SW, Courcoulas AP, Stylopoulos N. Gut adaptation after gastric bypass in humans reveals metabolically significant shift in fuel metabolism. Obesity (Silver Spring). 2023 Jan;31(1):49-61. doi: 10.1002/oby.23585. PMID 36541157
- [Background] Stefater-Richards MA, Panciotti C, Esteva V, Lerner M, Petty CR, Gourash WF, Courcoulas AP. Gastric bypass elicits persistent gut adaptation and unique diabetes remission-related metabolic gene regulation. Obesity (Silver Spring). 2024 Nov;32(11):2135-2148. doi: 10.1002/oby.24135. Epub 2024 Oct 15. PMID 39410706
- [Background] Courcoulas AP, Stefater MA, Shirley E, Gourash WF, Stylopoulos N. The Feasibility of Examining the Effects of Gastric Bypass Surgery on Intestinal Metabolism: Prospective, Longitudinal Mechanistic Clinical Trial. JMIR Res Protoc. 2019 Jan 24;8(1):e12459. doi: 10.2196/12459. PMID 30679147